CLINICAL TRIAL: NCT01128205
Title: Nationwide Assessment of Cardiovascular Risk Factors: Blood Pressure, Blood Lipid, and Blood Glucose, in Chinese Patients With Type 2 Diabetes, A Study of China Cardiometabolic Registries (CCMR)
Brief Title: Nationwide Assessment of Cardiovascular Risk Factors: in Chinese Patients With Type 2 Diabetes
Acronym: 3B
Status: Completed | Type: Observational
Sponsor: China Cardiometabolic Registries (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry); China Gerontological Society (Other); VitalStrategic Research Institute (Other)
Responsible Party: Li Nong Ji, MD, Peking Univeristy People's Hospital
Other Study IDs: CCMR-302-3B
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; cardiovascular risk factors; blood pressure; blood lipid; blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosed for 6 months or more

SUMMARY:
The objective of this study is to evaluate the level of control of cardiovascular disease risk factors, including blood pressure, blood lipid, and blood glucose, in out patients with type 2 DM in 6 representative regions in China: Northeast, North, East, South, Southwest and Northwest, measured by,

1. Proportion of patients reaching adequate control of blood glucose
2. Proportion of patients reaching adequate control of blood glucose and blood pressure, or blood glucose and blood lipid
3. Proportion of patients reaching adequate control of all 3Bs, i.e. blood glucose, blood pressure, and blood lipid.

DETAILED DESCRIPTION:
The prevalence of patients with diabetes mellitus (DM) worldwide has increased from 30 million in 1985 to 180 million at the present time. In China, the incidence of overweight, obesity, and DM has increased rapidly due to the significant change of diet and lifestyle resulted from rapid economic development. As estimated by International Diabetes Federation (IDF), the number of the patients with DM was about 39.8 million in China in 2007, and it is anticipated that the number would reach 59.3 million in 2025 [11]. At the same time there are a similar number of pre-diabetes patients with risk factors of cardiovascular diseases in China. DM and its associated microvascular and macrovascular complications could severely affects patients' quality of life and duration of survival and lead to significant increase in medical expenditure.

There have been a number of epidemiological surveys of diabetes conducted in other countries. However, there is little specific data available on the status of DM control and clinical outcomes of prevention and treatment of diabetic cardiovascular complications and other microvascular complications in China. This has made it difficult for clinicians to effectively make medical choices for patients with a variety of risk factors and complications.

This study is thus designed to assess the level of control of CVD risk factors, including blood pressure, blood lipid, and blood glucose, in outpatients with type 2 DM nation-wide across 6 representative regions in China: Northeast, North, East, South, Southwest and Northwest. The difference in clinical outcomes between the regions and between the three different tiers of hospitals, i.e. tier 3 (primary or teaching hospitals), tier 2 (secondary or city level hospitals), and tier 1 (community hospitals/health centers), will be made. The primary measurements include 1)Proportion of patients reaching adequate control of blood glucose (1B); 2)Proportion of patients reaching adequate control of blood glucose and blood pressure, or blood glucose and blood lipid (2B); and 3)Proportion of patients reaching adequate control of all 3Bs, i.e. blood glucose, blood pressure, and blood lipid. Other measurements include proportion of microvascular and macrovascular diabetic complications, DM treatment pattern and influence factors, physician prescribing behaviors, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with confirmed type 2 DM (According to ADA criteria) at least 6 month prior to the study visit;
2. At least 18 years or older;
3. Patients who are due and willing to receive a fasting blood testing within 7 days due to his/her underlying diseases, as determined by the investigator; or patients who have adequate blood test results obtained within 30 days;
4. Patients who are willing to sign consent form and are able to complete the questionnaires.

Exclusion Criteria:

1. Patients with type 1 DM;
2. Pregnant or breast feeding women;
3. Patients who are participating in any other clinical studies, including any questionnaire-based study, any interventional study (even diet/counseling based intervention), or any clinical trial in which any medication (including Chinese herbal medications) are administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese type 2 diabetic out-patients with diagnosis for 6 months or more
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The proportion adequate control of blood glucose, blood glucose and blood pressure or blood glucose and blood lipid, and blood glucose, blood pressure and blood lipid. | From the time of enrollment to within 30 day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — Peking University People's Hospital; Dayi Hu, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking Univresity People's Hospital, Beijing, China

REFERENCES:
- [Derived] Ji Q, Chai S, Zhang R, Li J, Zheng Y, Rajpathak S. Prevalence and co-prevalence of comorbidities among Chinese adult patients with type 2 diabetes mellitus: a cross-sectional, multicenter, retrospective, observational study based on 3B study database. Front Endocrinol (Lausanne). 2024 Jun 11;15:1362433. doi: 10.3389/fendo.2024.1362433. eCollection 2024. PMID 38919489
- [Derived] Cai X, Ji L. Generalizability of the Results of Cardiovascular Outcome Trials of Glucagon-Like Peptide 1 Receptor Agonists in Chinese Patients with Type 2 Diabetes Mellitus. Diabetes Ther. 2021 Jul;12(7):1861-1870. doi: 10.1007/s13300-021-01079-x. Epub 2021 May 28. PMID 34047959
- See also: Related Info — http://www.CCMRegistry.org